CLINICAL TRIAL: NCT03208569
Title: Treatment Optimization Regarding Anticholinergic Medications Potential Impact on Cognitive Test Performance
Brief Title: Anticholinergic Burden - Treatment Optimization
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Angelholm Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Studie ACB
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anticholinergics; Cognitive Function
Keywords: anticholinergic; alzheimer; cognition; MMSE; anticholinergic cognitive burden scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is increasing evidence that medications with anticholinergic effects may adversely impact cognitive function. Older adults are particularly sensitive to these effects due to age-related changes in pharmacokinetics and pharmacodynamics. The cumulative impact of taking one or more medications with anticholinergic properties is known as the anticholinergic burden. To quantify this burden, Boustani et al. (2008) developed the Anticholinergic Cognitive Burden (ACB) scale. The objective of this study is to examine whether optimizing pharmacotherapy concerning drugs with anticholinergic effects-identified by both the ACB scale and the newly developed Swe-ABS-can improve cognitive test performance among individuals attending a memory clinic. Anticholinergic drug use and cognitive performance will be assessed at baseline and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals aged ≥ 50 at the Memory Clinic, Hospital of Ängelholm
Sampling Method: Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 6 months
  Mini-Mental State Examination (MMSE). Range 0-30; maximum 30 indicating preserved cognitive functioning.
Cognitive function | 6 months
  Montreal Cognitive Assessment (MoCA). Range 0-30; maximum 30 indicating preserved cognitive functioning.
Cognitive function | 6 months
  Trail Making Test (TMT) - A. Assessing visual attention and processing speed. Age-dependent e.g, 65-74 years of age 33 ± 11 seconds. Trail Making Test (TMT) - B. Assessing executive function especially cognitive flexibiity. Age-dependent e.g, 65-74 years of age 85 ± 25 seconds.
Cognitive function | 6 months
  Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Neuropsychological test battery covering several cognitive domains. Age-dependent e.g, 70-79 years of age with education < 6 years: 12-16. High education: 8-12
Cognitive function | 6 months
  Symbol Digit Modalities Test (SDMT) Assessing attention, executive function and memory. Correctly identified symbols are recorded within a time frame of 90 seconds.
  Age-dependent e.g, 70-74 years of age with short education: 36. High education: 43
Cognitive function | 6 months
  A Quick Test of Cognitive Speed (AQT) Three moments, 1 color, 2 form and 3 color-form. Naming correctly as fast as possible.
Cognitive function | 6 months
  5x3 Memory Test A brief and structured memory test involving 15 concrete items grouped into five items on three subsequent sets.
  Scoring is based on immediate and delayed recall in a special scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Per Johansson, MD, PhD, Principal Investigator — Region Skåne
Locations (1):
- Specialistminnesmottagningen, Ängelholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rube T, Ecorcheville A, Londos E, Modig S, Johansson P. Development of the Swedish anticholinergic burden scale (Swe-ABS). BMC Geriatr. 2023 Aug 25;23(1):518. doi: 10.1186/s12877-023-04225-1. PMID 37626293
- See also: Article BMC Geriatr. 2023 Aug.25;23(1):518 — http://pubmed.ncbi.nlm.nih.gov/37626293/